CLINICAL TRIAL: NCT05865756
Title: Assessment of Radio(Chemo)Therapy-related Dysphagia in Head and Neck Cancer Patients Based on Cough-related Acoustic Features
Brief Title: Assessment of (Chemo)RT-related Dysphagia in HNC Patients Based on Cough-related Acoustic Features
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CE2762
Record Dates: First submitted 2023-04-17; First posted 2023-05-19 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-04

CONDITIONS: Head and Neck Cancer; Dysphagia
MeSH Terms: conditions — Head and Neck Neoplasms; Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: 40HNC patients in complete clinical remission (10 male/10 female adults & 10 male/10 female elderly) diagnosed with dysphagia treated with radiochemotherapy and selected three months after the end of treatment will be submitted to cough and voice analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cough and voice analysis in HNC patients (Other): Patients will undergo acoustic cough features analysis.
  Interventions: Other: Acoustic cough features analysis

INTERVENTIONS:
Other: Acoustic cough features analysis — Acoustic cough features analysis

SUMMARY:
To develop this objective and easily implementable assessment method of coughing based on acoustic features of voluntary and reflex coughs, there is a primary need in identifying and comparing acoustic cough features in healthy subjects and different disease-related coughs features. Cough is a common reason for seeking medical care. Chronic cough, defined as a cough that has lasted for longer that eight weeks, represents 10-38% of all referrals made to respiratory physicians [1-2]. Furthermore, between 60 and 80% of patients with chronic obstructivepulmonary disease (COPD) report cough. Following this pilot study comparing different populations, the applicability of the selected acoustic cough features should be examined in HNC patients with radiotherapy-induced dysphagia, Another frequent aspect of the clinical diagnostic examination of swallowing is perceptual analysis of voice quality immediately following deglutition. Changes in voice quality are assumed to provide information on the possible accumulation of saliva or food at the vocal folds level. It is reported that a change of voice may indicate laryngeal dysfunction or the presence of a foreign body at the laryngeal level [3] confirm that a normophonic voice after swallowing reflects a lack of aspiration-penetration. However, research shows that there is no strong correlation between aspiration and changes in perceptual voice quality (e.g. wet voice). A more reliable and easily implementable method could be detection of specific acoustic features of changes in voice quality.

DETAILED DESCRIPTION:
The ultimate goal of this study is to develop an innovative and non-invasive assessment method for dysphagia and aspiration in head and neck cancer (HNC) patients using acoustic features related to voluntary and/or reflex cough as biomarkers of dysphagia and/or aspiration in this population.

Additionally, the relationship between acoustic features and aerodynamic cough and acoustic voice parameters will be investigated, extending our insight in pathophysiology of dysphagia in this population.

To the investigators knowledge, no acoustic features of coughing and throat clearing in the frame of dysphagia have ever been explored. Regarding voice quality abnormalities, no acoustic parameters of reasonable evidence of dysphagia have been found.

ELIGIBILITY:
Inclusion criteria:

* HNC patients in complete clinical remission (10 male/10 female adults & 10 male/10 female elderly)
* Patients diagnosed with dysphagia (with evaluation by videofluoroscopy)
* Patients treated with radiochemotherapy and selected three months after the end of treatment.

Exclusion criteria:

-pulmonary diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
acoustic cough features in HNC patients as biomarkers for dysphagia/aspiration. | at least 3 months post-RT
  cough and voice analysis (using voice recording and frequencies obtained) of HNC patients post RT will be analysed to detect early diagnosis biomarkers for dysphagia/aspiration

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Jules Bordet, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Irwin RS, Curley FJ, French CL. Chronic cough. The spectrum and frequency of causes, key components of the diagnostic evaluation, and outcome of specific therapy. Am Rev Respir Dis. 1990 Mar;141(3):640-7. doi: 10.1164/ajrccm/141.3.640. PMID 2178528
- [Background] McGarvey LP, Heaney LG, Lawson JT, Johnston BT, Scally CM, Ennis M, Shepherd DR, MacMahon J. Evaluation and outcome of patients with chronic non-productive cough using a comprehensive diagnostic protocol. Thorax. 1998 Sep;53(9):738-43. doi: 10.1136/thx.53.9.738. PMID 10319055
- [Background] Waito A, Bailey GL, Molfenter SM, Zoratto DC, Steele CM. Voice-quality abnormalities as a sign of dysphagia: validation against acoustic and videofluoroscopic data. Dysphagia. 2011 Jun;26(2):125-34. doi: 10.1007/s00455-010-9282-4. Epub 2010 May 8. PMID 20454806